CLINICAL TRIAL: NCT02633579
Title: The Role of Induced Phase 3 Contractions in the Control of Hunger and Food Intake
Brief Title: Effect of the Motilin Receptor Agonist, Erythromycin, on Hunger and Food Intake; Study of Role of Cholinergic Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: ErythromycinHungerFoodIntake
Record Dates: First submitted 2015-11-02; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — erythromycin lactobionate; Erythromycin; Atropine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Erythromycin lactobionate (Active Comparator): 40 mg erythromycin lactobionate was administered over a 20 min period in a volume of 100 ml sodium chloride 0.9 %
  Interventions: Drug: erythromycin lactobionate
- Erythromycin lactobionate with atropine (Active Comparator): 40 mg erythromycin lactobionate was administered over a 20 min period in a volume of 100 ml sodium chloride 0.9 %; Atropine sulfate was given as an i.v. bolus (15 µg/kg) followed by a continuous infusion of 15 µg/kg/h over 30 min
  Interventions: Drug: Erythromycin with atropine
- Atropine (Placebo Comparator): Atropine sulfate was given as an i.v. bolus (15 µg/kg) followed by a continuous infusion of 15 µg/kg/h over 30 min.
  Infusion of saline as a placebo for erythromycin was administered over a 20 min period in a volume of 100 ml sodium chloride 0.9 %
  Interventions: Drug: Atropine
- Placebo (Placebo Comparator): Infusion of saline was administered over a 20 min period in a volume of 100 ml sodium chloride 0.9 %; also placebo for atropine was given as an i.v. bolus of saline followed by a continuous infusion over 30 min
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: erythromycin lactobionate — intravenous administration of erythromycin
  Other Names: Erythromycin
  Arms: Erythromycin lactobionate
Drug: Atropine — intravenous administration of atropine
  Arms: Atropine
Drug: Erythromycin with atropine — intravenous administration of erythromycin with saline
  Arms: Erythromycin lactobionate with atropine
Drug: Saline — intravenous administration of saline
  Other Names: Control
  Arms: Placebo

SUMMARY:
In this study, the investigators will evaluate if the food intake associated with the infusion of erythromycin is caused by the phase 3 contractions or by another yet unknown effect of erythromycin. To obtain this the investigators will use atropine, a muscarinic receptor antagonist, to inhibit the formation of contractions induced by a low dose of erythromycin

DETAILED DESCRIPTION:
The role of induced phase 3 contractions in the control of hunger and food intake

1. Background In between meals the motor activity of the upper gastrointestinal tract is characterized by a cyclical pattern of contractions that consists of 3 phases: maximal contractile activity originating in the stomach and migrating down the small intestine (phase 3), followed by a phase of motor quiescence (phase 1) and a phase of progressively increasing motor activity (phase 2). In 1975 Itoh et. al. linked the phase 3 contractions of the migrating motor complex (MMC) to hunger sensations, by increasing the hunger sensations through exogenously administered motilin. The investigators previously demonstrated that phase 3 is associated with a 'hunger pang'. The trigger for the phase 3 initiation is unclear, but the gut hormones ghrelin and motilin are presumed to play a role. If either of these substances are administered intravenously, they induce a premature phase 3 in humans.

   In previous studies, 'hunger pangs' could objectively be detected as peaks in subjective hunger ratings on a visual analog scale (VAS) using a custom made algorithm. A close association between phase 3 contractions of gastric origin and hunger peaks was observed and spontaneous food intake was also found to be associated with hunger peaks. By inducing phase 3 contractions through the administration of IV erythromycin, the time of food intake could be manipulated.

   In a new study the investigators will evaluate if the food intake associated with the infusion of erythromycin is caused by the phase 3 contractions or by another yet unknown effect of erythromycin. To obtain this the investigators will use atropine, a muscarinic receptor antagonist, to inhibit the formation of contractions induced by a low dose of erythromycin. Since food intake is no longer a pure physiological act to still hunger sensations, it has obtained a social and emotional status in modern times where palatable food is abundant, the relationship of the subject towards food using multiple questionnaires will also be evaluated.
2. Aim To investigate whether contractions in the antrum are necessary to induce food intake with erythromycin or if erythromycin has a secondary effect to stimulate food intake.
3. Methodology 3.1. Subject selection Healthy volunteers will be recruited. See eligibility criteria for details

3.2. Questionnaires

Dutch eating behaviour questionnaire (DEBQ):

The DEBQ will be administered as a measure of dietary restraint and disinhibition. The DEBQ investigates three fields of behavioral eating: restrained eating, emotional eating and external eating.

Council of nutrition appetite questionnaire (CNAQ):

This questionnaire is an appetite-monitoring instrument developed by the Council for Nutritional Strategies in Long-Term Care.

Hospital Anxiety & Depression Scale (HAD):

This questionnaire will be used to exclude subjects with mood & anxiety disorders.

Power of food scale (PFS):

The PFS evaluates the psychological impact of living in an environment where palatable food is abundant.

3.3. Protocol Study design Gastric motility will be registered for 7h after an overnight fast (see below). During this period the volunteers are allowed to ingest a standardized liquid meal twice at time points of their choice. The volunteers are exposed to the liquid meal before the start of the experiment and the palatability of the meal is scored; this is done in a standardized way (same cup, temperature, duration, only smelling not tasting). The liquid meal is a low-caloric soup with a similar composition as the one used by Hjelland et. al. The volunteers are not aware that the investigators want to study the association between gastric motility, hunger and food intake; they receive the information that the investigators want to examine the effect of fasting on the motility of the stomach and hunger. During the experiment they will watch standardized movies with a neutral emotional content at standardized time points. They will rate hunger every 5 minutes and they will be offered the opportunity to drink the meal at a time point of their choice. At the start of the experiment two intravenous catheters will be placed in separate arms of the subject. During the entire study saline will be administered intravenously at a low rate to blind the subject towards the time of drug administration. The infusion bag will be positioned behind a curtain, in this way the time of drug administration will be blind for the subject. The administration of the drug, 40 mg of the motilin receptor agonist erythromycin lactobionate (Erythrocine; Abbott, Ottignies-Louvain-la-Neuve, Belgium), will be given in a randomized fashion at time point 90, 180, 270 or 360 min after the start of the study. An infusion of this macrolide antibiotic will be given at two of the above time points, one of these erythromycin infusions will be preceded by a 15 µg/kg IV bolus of atropine (Stellatropine; Pharmacobel, Brussels, Belgium) plus a 30 min infusion of 15 µg/kg/hr of atropine. The administration of atropine will be given 10 minutes before the infusion of erythromycin in the opposite arm of the erythromycin infusion. The arterial pulse frequency will be monitored continuously during the administration of atropine. If the start point of an infusion coincides with a spontaneous phase 3, then the infusion will be postponed for 15 min until the phase 3 is passed.

Manometry Recording of antroduodenal intraluminal pressures will be performed using a Manoscan® high resolution manometry catheter (outer diameter 4.2 mm, 36 channels spaced 1 cm apart). The catheter will be introduced via the nose and the position of the catheter, see figure 1, will be briefly checked by fluoroscopy (typically 5 seconds, never more than 25 seconds). This part will comply with the relevant guidelines of radioprotection and participants will be protected by a leaden shield that covers the lower abdomen, Personnel will carry a leaden jacket, will not be exposed to the primary beam and will wear dosimeters at all time. The catheter will be placed in such a way, that there are measuring points in the antrum and just distal to the pylorus to accurately record the migrating motor complex. The output of the manometry channels is recorded and monitored on-line via the ManoScan 360™ (Sierra Scientific Instruments, Los Angeles, CA). After an overnight fast, the manometry assembly will be introduced as described above and secured to the subject's nose with adhesive tape. The subjects will then be positioned in a comfortable sitting position with the knees bent (80°) and the trunk upright in a specifically designed bed.

Behavioural ratings At 5-minute intervals, volunteers will indicate scores for hunger and expected amount to eat on a 10cm VAS. Emotions will be scored at a 15-minute interval on an electronic grid mood scale.

ELIGIBILITY:
Inclusion criteria:

* Female or male subjects aged 18 to 60
* Subject is capable and willing to give informed consent
* Female volunteers of child bearing potential must use oral, injected or implanted hormonal methods of contraception

Exclusion criteria:

* Female volunteer is pregnant or breastfeeding
* Gastrointestinal diseases, major abdominal surgery
* Major psychiatric illnesses
* Volunteers that use drugs affecting the gastrointestinal tract or the central nervous system
* Allergy for macrolide antibiotics
* Allergy for atropine
* Severe heartburn
* Enlarged prostate
* Blockage of urinary tract
* Acute closed-angle glaucoma
* Myasthenia gravies
* Severe heart disease
* Thyrotoxicosis
* Fever
* Liver problems
* High blood pressure or fast heart rate
* Lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in hunger ratings from time of administration over 6 hours | 6 hours after intervention, assessment every 5 minutes
  visual analog scale

SECONDARY OUTCOMES:
Timing of food intake | 6 hours after intervention; up to 2 moments of food intake allowed
  decision to take a soup meal

REFERENCES:
- [Background] Szurszewski JH. A migrating electric complex of canine small intestine. Am J Physiol. 1969 Dec;217(6):1757-63. doi: 10.1152/ajplegacy.1969.217.6.1757. No abstract available. PMID 5353053
- [Background] Itoh Z. AI, Takeuchi S., Couch E. F., editor. Hunger contractions and motilin. 5th International Symposium on Gastrointestinal Motility; 1975; Herentals, Belgium.
- [Background] Tack J, Deloose E, Ang D, Scarpellini E, Vanuytsel T, Van Oudenhove L, Depoortere I. Motilin-induced gastric contractions signal hunger in man. Gut. 2016 Feb;65(2):214-24. doi: 10.1136/gutjnl-2014-308472. Epub 2014 Dec 24. PMID 25539673
- [Background] Scarpellini E. HN, D. Ang, P. Vanden Berghe, I. Depoortere, J. Tack. Role of upper gastrointestinal motility stimulation in the occurence of hunger peaks. Gastroenterology. 2009;136:A330
- [Background] Janssens J, Vantrappen G, Peeters TL. The activity front of the migrating motor complex of the human stomach but not of the small intestine is motilin-dependent. Regul Pept. 1983 Aug;6(4):363-9. doi: 10.1016/0167-0115(83)90265-3. PMID 6635258
- [Background] Tack J, Depoortere I, Bisschops R, Delporte C, Coulie B, Meulemans A, Janssens J, Peeters T. Influence of ghrelin on interdigestive gastrointestinal motility in humans. Gut. 2006 Mar;55(3):327-33. doi: 10.1136/gut.2004.060426. Epub 2005 Oct 10. PMID 16216827
- [Background] Coulie B, Tack J, Peeters T, Janssens J. Involvement of two different pathways in the motor effects of erythromycin on the gastric antrum in humans. Gut. 1998 Sep;43(3):395-400. doi: 10.1136/gut.43.3.395. PMID 9863486
- [Background] Bayer LM, Bauers CM, Kapp SR. Psychosocial aspects of nutritional support. Nurs Clin North Am. 1983 Mar;18(1):119-28. PMID 6403929
- [Background] Patel KA, Schlundt DG. Impact of moods and social context on eating behavior. Appetite. 2001 Apr;36(2):111-8. doi: 10.1006/appe.2000.0385. PMID 11237346
- [Background] van Strien T, Oosterveld P. The children's DEBQ for assessment of restrained, emotional, and external eating in 7- to 12-year-old children. Int J Eat Disord. 2008 Jan;41(1):72-81. doi: 10.1002/eat.20424. PMID 17634965
- [Background] Soetens B, Braet C, Van Vlierberghe L, Roets A. Resisting temptation: effects of exposure to a forbidden food on eating behaviour. Appetite. 2008 Jul;51(1):202-5. doi: 10.1016/j.appet.2008.01.007. Epub 2008 Feb 7. PMID 18342989
- [Background] Wilson MM, Thomas DR, Rubenstein LZ, Chibnall JT, Anderson S, Baxi A, Diebold MR, Morley JE. Appetite assessment: simple appetite questionnaire predicts weight loss in community-dwelling adults and nursing home residents. Am J Clin Nutr. 2005 Nov;82(5):1074-81. doi: 10.1093/ajcn/82.5.1074. PMID 16280441
- [Background] Lowe MR, Butryn ML, Didie ER, Annunziato RA, Thomas JG, Crerand CE, Ochner CN, Coletta MC, Bellace D, Wallaert M, Halford J. The Power of Food Scale. A new measure of the psychological influence of the food environment. Appetite. 2009 Aug;53(1):114-8. doi: 10.1016/j.appet.2009.05.016. Epub 2009 Jun 12. PMID 19500623
- [Background] Hjelland IE, Ofstad AP, Narvestad JK, Berstad A, Hausken T. Drink tests in functional dyspepsia: which drink is best? Scand J Gastroenterol. 2004 Oct;39(10):933-7. doi: 10.1080/00365520410003344. PMID 15513330
- [Derived] Deloose E, Vos R, Janssen P, Van den Bergh O, Van Oudenhove L, Depoortere I, Tack J. The motilin receptor agonist erythromycin stimulates hunger and food intake through a cholinergic pathway. Am J Clin Nutr. 2016 Mar;103(3):730-7. doi: 10.3945/ajcn.115.113456. Epub 2016 Jan 27. PMID 26817505